CLINICAL TRIAL: NCT06185088
Title: Michigan ENdoluminal Distraction Device (MENDD) Tolerance Assessment Study
Brief Title: MENDD Tolerance Assessment Study
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Initial PI departed institution.
Sponsor: University of Michigan (Other)
Responsible Party: Principal Investigator, Meghan A. Arnold, MD, Clinical Associate Professor, University of Michigan
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: HUM00208413
Record Dates: First submitted 2023-12-14; First posted 2023-12-29 (Actual); Results first posted 2024-10-03 (Actual); Last update posted 2024-10-03 (Actual); Status verified 2024-09

CONDITIONS: Short Bowel Syndrome
MeSH Terms: conditions — Short Bowel Syndrome

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: Yes

ARMS (1):
- Participants with Ostomies (Other): Patients who have ostomies, and who are already undergoing a minor procedure for routine health screening or other health matters as standard of care.
  Interventions: Device: Coda® Balloon Catheters; Device: Double Balloon Endoscope (DBE)

INTERVENTIONS:
Device: Coda® Balloon Catheters — A balloon device that will be introduced into participants' intestine over a guide wire to test the radial stretch of the small bowel.
Device: Double Balloon Endoscope (DBE) — A balloon device that will be introduced retrograde through the ileostomy and the inter-balloon distance will be increased causing stretch on the intestine to test longitudinal stretch. The DBE will only be used if a participant tolerated the Coda® Balloon Catheter intervention.

SUMMARY:
This study will utilize approved devices in an off-label manner to create forces required to induce intestinal lengthening. Radial and longitudinal forces are both required, and two devices will be used to create forces in order to test tolerability of said forces. This is to provide evidence that humans could tolerate the forces produced by a proposed commercially built device.

This study will test the hypothesis that radial and longitudinal forces necessary to produce enterogenesis will cause low levels of discomfort in healthy adults. Approved devices will be utilized in an off-label manner to reproduce forces similar to our novel medical device which is designed to treat short bowel syndrome (SBS).

This trial will not be testing a treatment for SBS, and individuals with SBS are ineligible for recruitment.

ELIGIBILITY:
Inclusion Criteria:

* Existing Ileostomy older than 6 weeks Undergoing any existing procedure in endoscopy suite or operating room.

Exclusion Criteria:

* Inflammatory bowel disease of small bowel Pregnant Short bowel syndrome Bleeding disorder Chronic pain disorder Individuals taking chronic pain medications including prescriptions, cannabinoids or over the counter.

Individuals taking pain medications at the time of the procedure Cognitive Impairment to the extent that the questionnaire cannot be completed

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 1 (Actual)
Dates: Start 2023-03-06 (Actual); Primary Completion 2023-06-06 (Actual); Study Completion 2023-06-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Meghan A Arnold, MD, Principal Investigator — University of Michigan
Locations (1):
- Michigan Medicine, Ann Arbor, Michigan, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Participants With Ostomies
Started | 1
Completed | 1
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Participants With Ostomies
Number analyzed (Participants) | 1
Age, Customized [Count of Participants; unit: Participants]
  18 years to 99 years | 1
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1
  Male | 0
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0
  Not Hispanic or Latino | 0
  Unknown or Not Reported | 1
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 0
  More than one race | 0
  Unknown or Not Reported | 1
Region of Enrollment [Number; unit: participants]
  United States | 1

OUTCOME MEASURES:

1. Primary Outcome: Discomfort as Assessed by Visual Analog Scale (VAS) for Radial Stretch
Description: Participant discomfort will be assessed using VAS during radial stretch. The VAS is a scale ranging from 0 (no pain) to 10 (maximum pain).
Time Frame: 1-2 Minutes
Population: Because only one participant was involved in the entire trial, showing data could violate privacy interests.
Arm/Group | Participants With Ostomies
Number analyzed (Participants) | 0

2. Secondary Outcome: Discomfort as Assessed by Visual Analog Scale for Longitudinal Stretch
Description: Participant discomfort will be assessed using VAS during longitudinal stretch. The VAS is a scale ranging from 0 (no pain) to 10 (maximum pain).
Time Frame: Approximately 1 minute
Population: Because only one participant was involved in the entire trial, showing data could violate privacy interests.
Arm/Group | Participants With Ostomies
Number analyzed (Participants) | 0

ADVERSE EVENTS:
Time Frame: 30 days
Description: Because only one participant was involved in the entire trial, showing data could violate privacy interests.
Arm/Group | Participants With Ostomies
All-Cause Mortality (participants affected / at risk) | 0/0
Serious Adverse Events (participants affected / at risk) | 0/0
Other Adverse Events (participants affected / at risk) | 0/0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol (2023-10-04): https://cdn.clinicaltrials.gov/large-docs/88/NCT06185088/Prot_000.pdf